CLINICAL TRIAL: NCT04002583
Title: A Prospective Study Evaluating the Use of 48-hour Ambulatory EEG Monitoring in Early Onset Alzheimer's Disease
Brief Title: 48-hour Ambulatory EEG Monitoring in Early Onset Alzheimer's Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Neill R. Graff-Radford, M.D., Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 19-003078
Record Dates: First submitted 2019-06-27; First posted 2019-06-28 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Early Onset Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Early-onset Alzheimer's disease (EOAD) subjects (Experimental): Subjects with mild cognitive impairment due to EOAD will undergo a 48 hour computer assisted ambulatory electroencephalogram
  Interventions: Diagnostic Test: Computer assisted ambulatory electroencephalogram

INTERVENTIONS:
Diagnostic Test: Computer assisted ambulatory electroencephalogram — A portable 16 channel CAA-EEG is used to detect epileptiform abnormalities in a 48 hour ambulatory electroencephalogram (EEG)
  Other Names: CAA-EEG

SUMMARY:
Researchers are trying to determine the frequency of seizures and epilepsy in patients with Early-onset Alzheimer's disease (EOAD) using a 48-hour computer assisted ambulatory electroencephalogram.

ELIGIBILITY:
Inclusion criteria for EOAD patients will be recruited from the LEADS trial with the following:

* 40 to 64 years of age
* Meets NIA-AA criteria for mild cognitive impairment (MCI) due to AD or probable AD dementia.
* Have a global CDR score of ≤ 1.0
* Have capacity to provide informed consent (ICF) or has a legal authorized representative or guardian who provides IC.
* Amyloid positive status (PET scan with evidence of elevated amyloid)
* Must have a study partner (informant) who spends a minimum average of 10 hours per week with the participant (e.g., family member, significant other, friend, and caregiver) who is generally aware of the participants' daily activities and can provide information about the participant's cognitive and functional performance. If the participant does not have a study partner who spends 10 face-to-face hours per week, other arrangements for identifying a viable study partner will be granted on a case-by-case basis by the Site PI.
* Not pregnant or lactating. Women must be two years post-menopausal, be surgically sterile, or have a negative pregnancy test prior to each PET scan
* Fluent in English.

Exclusion Criteria:

* Meets core clinical criteria for non-AD dementia.
* Two or more first degree relatives with a history of EOAD suggestive of autosomal dominant transmission, unless known pathogenic mutations in APP, PSEN1, PSEN2 have been excluded.
* Known mutation in an ADAD gene (APP, PSEN1, PSEN2) or other autosomal dominant genes associated with other neurodegenerative disorders.
* MRI scans with evidence of infection or focal lesions, cortical strokes, multiple lacunes (single lacune is allowable unless it meets criteria for strategic lacune affecting cognition)
* Any significant systemic illness or unstable medical condition, which could lead to difficulty complying with the protocol (at the discretion of the Site PI)
* Medical history of a brain disorder other than the disorder causing dementia except for headache.
* Deemed ineligible by the Site PI for any other reason.

Ages: 40 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-02-19 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Electrographic seizures: Number of subjects with electrographic seizures | 48 hours
  Number of subjects with electrographic seizures in 48 hours on computer assisted ambulatory EEG

CONTACTS AND LOCATIONS:
Overall Officials: Neill Graff-Radford, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials